CLINICAL TRIAL: NCT06061861
Title: Kaiser Permanente Evaluating Nutritional Interventions in Food-Insecure High-Risk Adults (KP ENRICH) Study
Brief Title: Kaiser Permanente Evaluating Nutritional Interventions in Food-Insecure High-Risk Adults Study
Acronym: KP ENRICH
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2112426
Record Dates: First submitted 2023-09-12; First posted 2023-09-29 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Financial Support

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Financial Support and Free Delivery (Experimental): The intervention group will receive monthly financial support for healthy food items along with free home delivery through the Instacart platform.
  Interventions: Other: Financial support for healthy foods and free home delivery
- Free Delivery (Experimental): The control group will receive only free home delivery through the Instacart platform.
  Interventions: Other: Free home delivery

INTERVENTIONS:
Other: Financial support for healthy foods and free home delivery — Participants will receive monetary support to spend on healthy food items (e.g., vegetables and fruit) through the Instacart platform for a duration of 6 months and have home delivery and service fees waived for 4 orders per month through the Instacart platform for a duration of 6 months.
  Arms: Financial Support and Free Delivery
Other: Free home delivery — Participants will have home delivery and service fees waived for 4 orders per month through the Instacart platform for a duration of 6 months.
  Arms: Free Delivery

SUMMARY:
The goal of this randomized controlled trial is to compare the effect of receiving 6 months of monetary support for healthy food through a food delivery platform on change in glycosylated hemoglobin (HbA1c) levels among adults with type 2 diabetes mellitus with glycemic control that is above target level.

The main study aims are to:

1. To evaluate whether providing monthly financial support for home-delivered healthy food vs. only free food delivery through the Instacart platform reduces glycosylated hemoglobin levels within 6 months among Medi-Cal-insured Kaiser Permanente adult members with diabetes mellitus and suboptimal glycemic control.
2. To evaluate whether providing monthly financial support for home-delivered healthy food vs. only free food delivery through the Instacart platform reduces medical resource utilization within 6 months among Medi-Cal-insured Kaiser Permanente adult members with diabetes mellitus and suboptimal glycemic control.

DETAILED DESCRIPTION:
Eligible Kaiser Permanente adult members will be randomized to one of two groups:

1. Intervention arm, in which subjects will receive 6 months of monetary support (with up to 4 free home deliveries and no service fees) through the Instacart platform to select and receive healthy foods (e.g., vegetables and fruit).
2. Control arm, in which subjects will receive 6 months of free home deliveries and no service fees for up to 4 deliveries each month through the Instacart platform.

Glycosylated hemoglobin level will be assessed at baseline and at 6 months after enrollment. Medical resource utilization will be evaluated at 3 months, 6 months, and 12 months after enrollment. Patient-reported outcomes (i.e., diabetes quality of life, nutrition security, dietary habits, social needs, and food security) will also be assessed at baseline, 6 months, and 12 months after enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥18 years old at enrollment
* Active membership in Kaiser Permanente with Medi-Cal insurance and no additional private or commercial insurance
* Diagnosis of Type II diabetes mellitus (not including Type I diabetes mellitus or gestational diabetes mellitus)
* At least 2 outpatient glycosylated hemoglobin measures ≥7.5% in the prior 18 months
* Current access to the internet via computer or mobile device
* No interpreter needed

Exclusion Criteria:

* Advanced or end-stage kidney disease (estimated glomerular filtration rate ≤15 ml/min/1.73m^2 or receiving outpatient dialysis or having a prior kidney transplant)
* Known pregnancy at time of identification

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1007 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-12-27 (Actual); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
6-month change in glycosylated hemoglobin level | 6 months after enrollment
  Baseline glycosylated hemoglobin will be ascertained using routine laboratory tests in the electronic health record prior to enrollment. Participants will complete glycosylated hemoglobin testing 6 months after enrollment.

SECONDARY OUTCOMES:
12-month change in glycosylated hemoglobin level | 12 months after enrollment
  Glycosylated hemoglobin will be ascertained using routine laboratory tests in the electronic health record at 12 months after enrollment.
Percentage of participants with glycosylated hemoglobin <7.5% | 6- and 12-months after enrollment
  Baseline glycosylated hemoglobin will be ascertained using routine laboratory tests in the electronic health record prior to enrollment. Participants will complete glycosylated hemoglobin tests 6 months after enrollment. 12-month glycosylated hemoglobin level will be ascertained using routine laboratory tests in the electronic health record.
All-cause hospitalizations or emergency department visits | 3-, 6-, and 12-months after enrollment
  Occurrence of hospitalization or emergency department visit for any reason within 12 months after enrollment.
Change in self-reported level of food security | 6- and 12-months after enrollment
  Participants will answer 10 questions about their food security using the USDA adult food security module. Affirmative responses to questions will be assigned 1 point in the food security scale (out of 10). Participants will be classified as being food secure (0-2 points) or food insecure (3-10 points).
Change in self-reported level of nutrition security | 6- and 12-months after enrollment
  Participants will be asked about their level of difficulty in accessing healthy food on a 5-point Likert scale. Participants will also be asked 13 questions on reasons for not eating healthy food, with each question scored from 0-2 (Never, Sometimes, Often true). Lower scores indicate higher nutrition security.
Change in self-reported dietary habits | 6- and 12-months after enrollment
  Participants will be asked 8 questions to examine their consumption of fast food, fruits, vegetables, legumes, nuts, dairy, seafood, sweets, and sugar-sweetened beverages over the past month.
Change in self-reported diabetes-related quality of life | 6- and 12-months after enrollment
  Participants will answer 13 questions about their diabetes-related quality of life, each on a 5-point Likert scale. Scores range from 13-65, with higher scores indicating lower diabetes-related quality of life.
Change in self-reported readiness to change | 6- and 12-months after enrollment
  Participants will be asked about their readiness to change their dietary habits to manage their diabetes on a 5-point Likert scale.

CONTACTS AND LOCATIONS:
Overall Officials: Claudia L Nau, PhD, Principal Investigator — Kaiser Permanente; Richard Grant, MD, MPH, Principal Investigator — Kaiser Permanente
Locations (2):
- United States (2):
  - Kaiser Permanente Southern California Department of Research & Evaluation, Pasadena, California
  - Kaiser Permanente Northern California Division of Research, Pleasanton, California

IPD SHARING:
Plan to Share IPD: No